CLINICAL TRIAL: NCT03442426
Title: Transforming Primary Care for Older Canadians Living With Frailty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Dalhousie University (Other); University of Calgary (Other); University of British Columbia (Other); Laval University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ORE22446
Record Dates: First submitted 2017-12-04; First posted 2018-02-22 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Frail Elderly Syndrome
Keywords: Primary Health Care; Frail Elderly; Qualitative Methods; Quantitative Methods; Cost-Benefit Analysis; Patient Participation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: We have proposed a strong quasi-experimental alternative with inclusion of a usual care group of patients prior to initiation of the intervention. Specifically, our study will use a quasi-experimental control group design with pre-test and post-test. Our control group will receive usual care, and the intervention group will receive the proposed intervention (screening, care coordination and individual care plans, engagement in decision making, and technology support). The usual care group will be followed for 6 months after study entry (baseline period). Once completed, the intervention will be implemented and recruitment for the intervention group will begin. The intervention group will also be followed for 6 months after study entry (intervention period). We will be able to compare the intervention group with the usual care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Cohort (Experimental): Integrated model of primary care
  Interventions: Other: Integrated model of primary care

INTERVENTIONS:
Other: Integrated model of primary care — Intervention includes: 1) consistent risk screening and assessment; 2) care coordination and system navigation; 3) patient/caregiver engagement and shared decision-making; and 4) enabling technology supports.

SUMMARY:
It is well known that older Canadians are high users of health care services. What is less well known is that the health care system is not well-designed to meet the needs of those who use it most. Older persons look to their primary care practitioners to assess their needs and coordinate their care. Unfortunately, the health concerns of older persons are often missed in too-short office visits. They may need care from a variety of providers and services, but this care is often not well-coordinated. Older persons and their caregivers are the experts in their own needs and preferences, but often do not have a chance to participate fully in treatment decisions or care planning. As a result, they may have health problems that are not properly assessed, managed or treated resulting in poorer health, as well as preventable and expensive emergency department visits and hospital stays.

Improving the health of older Canadians means identifying health problems early. It means providing timely supports so that manageable concerns do not spiral out of control. And, above all, it means helping health care providers actively engage older patients and their family caregivers as partners in care. Patients want to make informed choices about their health and the care they receive, based on their personal values, preferences and goals, and informed by available evidence.

Nine primary care clinics in three provinces (Quebec, Ontario, Alberta) will use a quick screening tool to identify older patients who are at risk of becoming frail. This will help initiate referral to health care or support services where necessary. Innovative technology will be used to streamline the referral process and help assist older adults in decision-making about their care.

With support from the Canadian Frailty Network (CFN, formerly TVN), researchers, collaborators, health care providers and older adults from across Canada will work together to transform primary health care for frail elderly Canadians.

DETAILED DESCRIPTION:
The team will be implementing evidence-based and tested interventions as a coherent strategy to enhance primary health care for older adults, working collaboratively with study sites, older adults, and other stakeholders to develop a scalable and sustainable model. The investigators aim to develop the capacity of primary health care teams to identify, assess, and support older adults (70+) who are frail, and to delay or prevent decline for those at lower risk. The project will support patient/caregiver engagement, and stronger care coordination and integration with other health and social services. The primary research question is: compared to usual care in primary care settings, does the proposed model improve health, social and economic outcomes for frail and at-risk older Canadians (aged 70+)? The investigators hypothesize that older adults will benefit from screening, active engagement in care planning, and appropriate referrals to services earlier in their care trajectories. In addition to improving health outcomes and quality of life for patients, more proactive interventions can reduce costly emergency department visits and unplanned hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* older adults age 70+ who attend the primary care clinic, speak and understand English language

Exclusion Criteria:

* older adults less than 70 years of age, patients who don't not speak/understand English, patients living in long-term care, patients not rostered for 6 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 695 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Assessing change in 'Care for Chronic Conditions' scores | The tool will be used at 4 time points: at baseline recruitment (B1), then 6 months later (B2), then 6 months later following intervention implementation (I1), and 6 months later (I2). Scores will be compared pre and post.
  This tools measures specific items related to the Chronic Care Model, and reports on patient experience with the system. There are 5 sub scales (patient activation, delivery system, goal setting, problem solving and coordination) and 26-items. This tool has been validated.

SECONDARY OUTCOMES:
Assessing change in 5-Level EQ-5D questionnaire | The tool will be used at 4 time points: at baseline recruitment (B1), then 6 months later (B2), then 6 months later following intervention implementation (I1), and 6 months later (I2). Scores will be compared pre and post.
  This tool measures health-related quality of life. The tool is comprised of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression).
Assessing change in the Canadian Institute for Health Information Primary Care Provider Survey | This tool will be used at two time points. Once at baseline (B1) and again at the end of the study (2.5 years later) post implementation (I2). All providers involved in the work will completed the tool.
  This survey addresses team function, involvement in governance, use of information technology and scope of practice.
Assessing Healthcare Utilization across different time points | The tool will be used at 4 time points: at baseline recruitment (B1), then 6 months later (B2), then 6 months later following intervention implementation (I1), and 6 months later (I2). Scores will be compared pre and post.
  Self-reported health care utilization data including hospital admissions; emergency department visits, home care services; specialist visits and primary care visits.

OTHER OUTCOMES:
Assessing change in Goal Attainment Scaling (GAS) | GAS will be completed with a small sub-set of participants during qualitative interviews at baseline recruitment (B1), then 6 months later (B2), then 6 months later following intervention implementation (I1), and 6 months later (I2).
  GAS is an individualized, client-centred goal-setting and measurement approach that can accommodate a client's individual wishes, values and preferences. Goals are scaled on a five-point rating scale from -2 (much less than expected) to +2 (much better than expected). The GAS formula translates the total GAS score into a standardized score, with a score of 50 representing overall goal attainment.
Assessing change in Canadian Institute for Health Information Primary Care Organizational Survey | This tool will be used at two time points. Once at baseline (B1) and again at the end of the study (2.5 years later) post implementation (I2).All providers involved in the work will completed the tool.
  This survey is usually completed by a manager or director of the primary care site. The survey covers many domains such as human resources, accessibility, coordination, quality improvement, and system integration.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stolee, Dr., Principal Investigator — University of Waterloo
Locations (3):
- Canada (3):
  - Alberta PCNs, Calgary, Alberta
  - Quebec Primary Care, Québec, Quebec
  - Ontario Primary Care, Waterloo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sims-Gould J, Elliott J, Tong CE, Giguere A, Mallinson S, Stolee P. A national intervention to support frail older adults in primary care: a protocol for an adapted implementation framework. BMC Geriatr. 2021 Aug 4;21(1):453. doi: 10.1186/s12877-021-02395-4. PMID 34348660
- [Derived] Stolee P, Elliott J, Giguere AM, Mallinson S, Rockwood K, Sims Gould J, Baker R, Boscart V, Burns C, Byrne K, Carson J, Cook RJ, Costa AP, Giosa J, Grindrod K, Hajizadeh M, Hanson HM, Hastings S, Heckman G, Holroyd-Leduc J, Isaranuwatchai W, Kuspinar A, Meyer S, McMurray J, Puchyr P, Puchyr P, Theou O, Witteman H. Transforming primary care for older Canadians living with frailty: mixed methods study protocol for a complex primary care intervention. BMJ Open. 2021 May 13;11(5):e042911. doi: 10.1136/bmjopen-2020-042911. PMID 33986044